CLINICAL TRIAL: NCT00291824
Title: A Randomized Controlled Trial of the Effects and Expense of a Primary and Secondary Cardiovascular Risk Reduction Clinic in Primary Care
Brief Title: Cardiovascular Lifestyle Study: Effects and Expense of a Cardiovascular Risk Reduction Clinic in Primary Care
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Caroline Medical Group (Other)
Collaborators: Health Canada (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PHCTF G03-02656
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2006-02-15 (Estimated); Status verified 2006-02

CONDITIONS: Hypertension; Hyperlipidemia; Hyperglycemia; Cardiovascular Disease; Smoking
Keywords: Cardiovascular risks; Motivational interviewing; Behavior change; Primary care setting
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Hyperglycemia; Cardiovascular Diseases; Smoking | interventions — Heart Disease Risk Factors

INTERVENTIONS:
Behavioral: Cardiovascular risk factors and willingness to change

SUMMARY:
The purpose of this trial is to study the effects on risk reduction and expense of 3 approaches to the care of people with cardiovascular risk factors in a naturalistic primary care environment.

DETAILED DESCRIPTION:
Background: Uncontrolled hypertension, hyperlipidemia, hyperglycemia, smoking and other cardiovascular risks remain at epidemic proportions despite known efficacious treatments. Issues of both provider and patient behavioral non-adherence to guidelines and therapeutic regimes, respectively, are key factors in non-control. Few interventions aimed at reducing cardiovascular risk factors are based on sound theories of behavior change.

Objective: To assess the effectiveness and expense of three approaches to the care of persons with known risks for cardiovascular disease. The three treatment approaches are usual care, usual care plus nurse telephone calls, and usual care plus clinic visits to a nurse and/or physician.

Design: Patients will be randomized to a 1) specialized proactive, and holistic cardiovascular risk management clinic using principles of behavior change; 2) nurse telephone calls as an attention placebo, yet a low dose, health promotion intervention; and 3) usual primary care. A random sample of 670 patients with cardiovascular risks identified in the past five years will be selected. Patients will be excluded if they do not speak English, are cognitively impaired or live in a nursing home. Interview questionnaires will measure cardiovascular risk, intention to change, social support, depression, coping and health services use. In addition, patients will be required to give a blood sample to measure cholesterol and glucose levels. Patients will then be randomized to one of three treatment groups.

Significance: The expected findings of this study is that the cardiovascular clinic, with nurse and physician, will be most effective at reducing cardiovascular risk and will pay for itself by averting hospital and emergency use for cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* A random sample of all persons with visits to their primary care physician for cardiovascular risks in past year. Cognitively intact (mini-mental state) or living with a carer who is cognitively intact. All other co-morbidities

Exclusion Criteria:

* Presently in a nursing home or in-patient long-term care facility (already receiving medications and diets as prescribed). No available family/friend interpreter if non-English speaking.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 670
Dates: Start 2004-08; Study Completion 2006-02

PRIMARY OUTCOMES:
Current Interview or Chart
International classification of diseases
Characteristics/demographics (dob, gender, marital status, living arrangement, employment, culture, language, spiritual beliefs, concurrent diseases - number/type).
Cognition: 10 item short portable mental status questionnaire (SPMSQ)(Pfeiffer, 1975)
Number of MD visits for cardiovascular risk factor
Percentage change in cardiovascular risk scores over time.
Percentage of targeted weight and exercise goals achieved (blood pressure control, smoking cessation, weight control, cholesterol control, sugar control, exercise levels). (Grundy, et al, 1999)
Self efficacy scale (Lorig et al, 1996)
Social support - personal resource questionnaire 85 (Weinert & Brandt 1987).
Depression (MADRS)(Montgomery & Asberg 1979) (Montgomery et al 1985) (Browne, Steiner Roberts et al 2002).
Coping (Moos and Billings 1984)
Expenditures of health and social services (Browne et al 2001)
Calculate the number of Framingham points for each risk factor
Blood samples
Counselling
Education

SECONDARY OUTCOMES:
Motivational Interviewing
Behavior Change

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mills, MD CCFP, Principal Investigator — Caroline Medical Group
Locations (1):
- Caroline Medical Group, Burlington, Ontario, Canada